CLINICAL TRIAL: NCT01539824
Title: A Phase II, Single Arm, Investigative Study of IMM-101 in Combination With Radiation Induced Tumour Necrosis in Patients With Previously Treated Colorectal Cancer
Brief Title: A Study of IMM-101 in Combination With Radiation Induced Tumour Necrosis in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM-101-007; 2011-003958-85 (EudraCT Number)
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IMM-101; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMM-101 plus SBRT (Experimental): The treatment regimen with IMM-101 (Mycobacterium obuense) will be every 2 weeks for the first three doses with the last of these doses being on the same day as the radiotherapy by CyberKnife treatment on a liver lesion targeted by the Principal Investigator. Following a rest of 4 weeks, patients will again receive IMM-101 every 2 weeks for the next 3 doses followed by a further 4 weeks rest. Thereafter, IMM-101 will be given at 4 week intervals for up to 12 months or until patient withdrawal for any reason
  Interventions: Biological: Mycobacterium obuense; Radiation: SBRT

INTERVENTIONS:
Biological: Mycobacterium obuense — IMM-101 is a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
  Other Names: IMM-101
Radiation: SBRT — The CyberKnife system is normally used for the treatment of cancerous tumours in cases where the type and position of the tumour and the condition of the patient indicate that treatment may be curative. In this study, the CyberKnife is being used in an experimental way to deliver a targeted dose of stereotactic body radiation with extreme accuracy in order to damage a single tumour growth (metastasis) in the liver.
  Other Names: stereotactic body radiation; CyberKnife

SUMMARY:
The purpose of this study is to investigate the safety and effects of IMM 101 in combination with a single targeted dose of radiation in patients with metastatic colorectal cancer in whom chemotherapy or other treatment has not been effective. Administration of radiation (using the CyberKnife) to the target tumour growth in the liver results in the release of tumour material. IMM-101 may help the immune system to react to the tumour material released from the damaged tumour, and so have a beneficial effect in slowing down the rate of growth of other tumour growths in the liver and other organs.

DETAILED DESCRIPTION:
Radiotherapy given in standard fractionation regimes leads to cell death by causing double stranded DNA breaks via production of oxygen free radicals. At the very high doses of stereotactic body radiotherapy (SBRT) administered with extreme accuracy in a single fraction by the CyberKnife system, there is induction of tumour necrosis due to endothelial cell damage and vascular collapse, cell membrane breakdown, and the release of cellular material and tumour antigens into the circulation, in addition to DNA strand breaks. It is hypothesised that the combination of modulation of the body's immune responses in the presence of an increased exposure to tumour antigen will provide sufficient induction of the immune system to suppress tumour growth.

ELIGIBILITY:
Inclusion criteria:

Male or female; aged ≥ 18 years. Histologically confirmed colorectal adenocarcinoma. Documented evidence of disease progression following at least one line of chemotherapy.

No further standard chemotherapy options available have refused further chemotherapy.

Metastatic lesions in at least two sites in the liver (+/- other sites) suitable for bidimensional and volumetric evaluation by CT scan.

World Health Organization (WHO) performance status of 0-2. Cockcroft calculated Glomerular Filtration Rate of > 40mL/min at screening. Life expectancy, in the opinion of the Investigator, of > 3 months from screening.

Exclusion Criteria:

Evidence of central nervous system metastasis. Severe, active uncontrolled infection requiring systemic antibiotics, antiviral or antifungal treatments.

Any previous or concurrent malignancy, except adequately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin and/or non-melanoma skin cancer, or if previous malignancy was more than 5 years earlier and there are no signs of recurrence.

Serum albumin < 30 g/L at screening. C-reactive protein (CRP) > 70 mg/L at screening. Transaminases (ALT or AST) > 5 X Upper Limit of Normal at screening. Bilirubin level > 2 X Upper Limit of Normal at screening. Radiotherapy in the 12 weeks before screening. Depot corticosteroid use in the 6 weeks before screening. Chronic use of any systemic corticosteroids (> 10 mg per day of prednisolone or equivalent for a period of 2 weeks or more) and/or immunosuppressant drugs (such as azathioprine, tacrolimus, cyclosporin) within the 2-week period before the first administration of study drug.

Woman of child-bearing potential who is not using an approved method of birth control Any investigational product administration in the 3 months before screening. Contraindication to CT scan, e.g., allergy to iodine based contrast medium. A surgical or medical condition which, in the judgement of the Investigator, might interfere with the activity of IMM-101, or with the performance of this study.

Any uncontrolled concomitant disease which, in the judgement of the Investigator, might interfere with the activity of IMM-101, or with the performance of this study.

History of serious adverse reaction or serious hypersensitivity to any drug that in the opinion of the Investigator may raise a safety concern.

Any previous treatment with IMM-101 or related mycobacterial immunotherapy (prior bacillus Calmette-Guerin (BCG) vaccination against Tuberculosis is allowed).

Known history of human immunodeficiency virus (HIV) or syphilis, current symptomatic Hepatitis B or C.

Unable or unwilling to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2014-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gaya, Principal Investigator — Leaders In Oncology Care, Harley St, London
Locations (2):
- United Kingdom (2):
  - HCA International, The Sarah Cannon Research Institute, London
  - The London Clinic, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IMM-101 Plus Stereotactic Body Radiation Therapy (SBRT): The treatment regimen with IMM-101 (Mycobacterium obuense) will be every 2 weeks for the first three doses with the last of these doses being on the same day as the radiotherapy by CyberKnife treatment on a liver lesion targeted by the Principal Investigator. Following a rest of 4 weeks, patients will again receive IMM-101 every 2 weeks for the next 3 doses followed by a further 4 weeks rest. Thereafter, IMM-101 will be given at 4 week intervals for up to 12 months or until patient withdrawal for any reason
  Mycobacterium obuense: IMM-101 is a suspension of heat-killed whole cell M. obuense in borate-buffered saline.
  SBRT: The CyberKnife system is normally used for the treatment of cancerous tumours in cases where the type and position of the tumour and the condition of the patient indicate that treatment may be curative. In this study, the CyberKnife is being used in an experimental way to deliver a targeted dose of stereotactic body radiation with extreme accuracy in order to damage a single tumour growth (metastasis) in the liver.
Period: Overall Study
Arm/Group | IMM-101 Plus Stereotactic Body Radiation Therapy (SBRT)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMM-101 Plus SBRT
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Disease Stabilisation Rate
Description: The disease stabilisation rate at 24 weeks defined as the proportion of patients with a complete response, partial response or stable disease in accordance with immune-related response criteria.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101 Plus SBRT
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Safety and Tolerability Profiles
Description: Safety and tolerability profiles as judged by:
  Local and systemic toxicities. Number, type and degree of toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) v4.0.
  Safety and tolerability are be monitored through the study by a Data Monitoring Committee (DMC)
Time Frame: 48 weeks
Population: All enrolled patients
Measure: Number; unit: Adverse event
Arm/Group | IMM-101 Plus SBRT
Number analyzed (Participants) | 12
Adverse event
  Serious adverse events (SAE) reported | 0
  Adverse events (AE) reported | 156

3. Secondary Outcome: Objective Response Rate
Description: Patients with an objective response were those who had a complete (CR) or partial response (PR), or stable disease(SD) based on CT scan findings, absence of clinical signs and symptoms of progression, did not withdraw due to disease progression prior to/at the Week 12/ 24 /36 / 48 assessment and were alive at the relevant assessment point
Time Frame: 12, 24, 36 and 48 weeks
Population: All enrolled patients who were still in follow up at each timepoint
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Population: All enrolled patients were included in the analysis population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 12
Participants
  Number of patients with objective response at Week 12 | 0
  Number of patients with objective response at Week 24 | 0
  Number of patients with objective response at Week 36 | 0
  Number of patients with objective response at Week 48 | 0

4. Secondary Outcome: Disease Stabilisation Rate
Description: Patients with disease stabilisation were those who had CR, PR, or SD based on CT scan findings, absence of clinical signs and symptoms of progression, did not withdraw due to disease progression prior to/at the Week 24, 36 or 48 assessment and were alive at the respective assessment.
Time Frame: 12, 36 and 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 12
Participants
  Number of patients with disease stabilisation at Week 12 | 0
  Number of patients with disease stabilisation at Week 36 | 0
  Number of patients with disease stabilisation at Week 48 | 0

5. Secondary Outcome: Overall Disease Stabilisation Rate
Description: The overall disease stabilisation rate was recorded as the percentage of patients with a CR, PR or SD as best overall response and was to be assessed at 12, 24 (primary time point), 36 and 48 weeks and overall.
Time Frame: 12, 36 and 48 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 12
Participants
  Overall disease stabilisation rate at Week 12 | 0
  Overall disease stabilisation rate at Week 36 | 0
  Overall disease stabilisation rate at Week 48 | 0

6. Secondary Outcome: Overall Response Rate
Description: The overall response rate will be recorded as the percentage of patients with a CR or PR as best overall response.
Time Frame: 12, 24, 36 and 48 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 12
Participants
  Overall response rate at Week 12 | 0
  Overall response rate at Week 24 | 0
  Overall response rate at Week 36 | 0
  Overall response rate at Week 48 | 0

7. Secondary Outcome: Survival
Description: The number of patients alive at 12, 24, 36 & 48 weeks. Patients without a date of death were to be censored at the date the patient was last known to be alive. The protocol made provision for patients to continue to be followed up and data to be collected, post study withdrawal.
Time Frame: 12, 24, 36 and 48 weeks
Population: One patient died during the study due to the AE of Jaundice (unrelated to IMM-101). The remaining 11 patients died after withdrawal from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 12
Participants
  Number of patients alive at 12 weeks | 10
  Number of patients alive at 24 weeks | 6
  Number of patients alive at 36 weeks | 3
  Number of patients alive at 48 weeks | 2

ADVERSE EVENTS:
Time Frame: From screening until end of study (up to 54 weeks)
Description: It was the responsibility of the investigator to report any directly observed AEs and AEs reported spontaneously by the patient, throughout the study after patient consent, and for IMM-101-related AEs, up to 30 days after the last study visit.
Arm/Group | Overall Study Population
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Population (N=12)
Fatigue (General disorders) | 7 (9)
Injection site reaction (General disorders) | 4 (13)
Peripheral odeama (General disorders) | 2 (5)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Influenza like symptoms (General disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Temperature intolerance (General disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 3 (3)
Gamma glutamyltransferase increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
RBC sedimentation rateincreased (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (2)
Blood urine present (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (2)
Carcinoembryonic antgen increased (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Urine ketone body present (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal psin (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
SCiatica (Nervous system disorders) | 1 (2)
Jaundice (Hepatobiliary disorders) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 1 (2)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Cardiac insufficiency (Cardiac disorders) | 1 (1)
Sinus tachtcardia (Cardiac disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The success criteria for the study as a whole, including progression to the second stage, were challenging. With hindsight, a larger sample size facilitating analysis of a less demanding, but still clinically meaningful, treatment effect might have been more appropriate and would be recommended for any future similar investigations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No